CLINICAL TRIAL: NCT07002788
Title: Comparison of Postoperative Analgesic Efficacy of Paravertebral Block and Serratus Anterior Plane Block in Patients Undergoing Video-assisted Thoracoscopic Surgery (VATS)
Brief Title: Comparison Paravertebral and Serratus Anterior Plane Block in Video-assisted Thoracoscopic Surgery.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Murat İzgi, assistant professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-24035
Record Dates: First submitted 2025-03-16; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer (NSCLC); Lung Adenocarcinoma; Video Assisted Thoracic Surgery (VATS)
Keywords: paravertebral block; serratus anterior plane block; lung cancer; video-assisted thoracoscopic surgery
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Bupivacaine; Morphine; Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paravertebral block (Active Comparator): Paravertebral block: After the patient is in the lateral decubitus position and the necessary antiseptic conditions are provided, the linear probe of the ultrasound will be placed between two transverse processes in the paramedian plane on the side to be operated on, and the transverse processes and the superior costotransverse ligament and pleura will be visualized at the level of the thoracic 6-7 vertebrae. The 22 gauge 50 mm needle will be advanced in-plane with ultrasonography until it passes the superior costotransverse ligament, and 20 ml of 0.5% bupivacaine hydrochloride will be injected while the needle tip is in the thoracic paravertebral area. The spread of the local anesthetic drug and the collapse movement of the pleura will be observed on ultrasonography.
  Interventions: Drug: Bupivacaine; Drug: Morphine; Drug: Paracetamol; Drug: Diklofenak Sodyum
- serratus anterior plane block (Active Comparator): In patients who will undergo serratus anterior plane block, after the necessary antiseptic conditions are provided in the lateral decubitus position, 30 ml of 0.25% bupivacaine hydrochloride will be injected into the anatomical neurofascial space between the serratus anterior and latissimus dorsalis muscle with a 10 cm long block needle in the mid-axillary line between the 4th and 5th ribs using the linear probe of the ultrasound.
  Interventions: Drug: Bupivacaine; Drug: Morphine; Drug: Paracetamol; Drug: Diklofenak Sodyum

INTERVENTIONS:
Drug: Bupivacaine — Used for regional anesthesia during VATS procedure (e.g., paravertebral or serratus anterior plane block)
  Other Names: Bupivakain
Drug: Morphine — Used for postoperative pain control via PCA device.
  Other Names: morfin
Drug: Paracetamol — Used as part of postoperative multimodal analgesia
  Other Names: Acetaminophen
Drug: Diklofenak Sodyum — Administered for postoperative pain management
  Other Names: NSAID

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) is a minimally invasive alternative to thoracotomy that emerged in the early 1990s, aiming to reduce surgical stress and postoperative pain. While VATS generally results in less pain than thoracotomy, patients may still experience significant discomfort. Effective pain control remains crucial in VATS to minimize postoperative complications, especially pulmonary and cardiac events, which can arise from inadequate ventilation and impaired sputum clearance due to pain.

Various strategies have been developed to manage postoperative pain, with multimodal approaches-combining regional or peripheral blocks with systemic analgesics such as NSAIDs and adjuvants-now considered standard. Among regional techniques, serratus anterior plane (SAP) block and thoracic paravertebral block (PVB) are commonly used. SAP block targets the thoracodorsal, long thoracic, and T2-T9 spinal nerves between the latissimus dorsi and serratus anterior muscles, providing effective anterolateral chest wall analgesia. PVB targets intercostal nerves within the paravertebral space and has shown superior pain control and improved lung function compared to systemic opioids or intrapleural local anesthetics.

At our center, both SAP and PVB are routinely used for postoperative analgesia in VATS procedures for patients with lung masses. Pain levels will be assessed using the Visual Analog Scale (VAS), a reliable tool for evaluating both acute and chronic pain, unaffected by age or gender.

This study aims to compare the effectiveness of SAP and PVB blocks in terms of postoperative pain, opioid requirements, and block-related complications in patients undergoing VATS under general anesthesia. The research is observational and will not alter routine clinical practices.

DETAILED DESCRIPTION:
The study is a single-center randomized single-blind prospective clinical study, and after patients with appropriate criteria are included in the study; they will be assigned to either the paravertebral block arm or the serratus anterior plane block arm of the study using an internet-based randomization program (randomizer.org). Patients will not know which arm of the study they are in, but researchers who will evaluate the treatment outcome will know which block was applied to which patient. Paravertebral block or serratus anterior plane block will be applied to the patients under general anesthesia after VATS according to the arm they are in. After the patients are taken to the room, non-invasive arterial blood pressure, electrocardiogram, and peripheral oxygen saturation monitoring will be performed before general anesthesia. This is the routine monitoring method applied before anesthesia application. Standard routine general anesthesia will be applied to the patients. No change will be made in the general anesthesia approach due to the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-64 who gave consent to participate in the study
* Patients between the ages of 65-90 who received a score of 24 or more from the mini mental test and gave consent to participate in the study
* ASA 1-3 patients

Exclusion Criteria:

* Those with neuropathy,
* Those with renal failure,
* Those with liver failure,
* Those with coagulopathy,
* Those with local anesthetic allergy,
* Those with infection in the area where the procedure will be performed,
* Those with congenital muscle absence in the area where the block will be performed
* Patients who did not give consent to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Scores (VAS) | Within the first 24 hours after surgery
  Pain assessment will be performed by Res. Asst. Dr. Rabia Çakmak at the 1st, 3rd, 6th, 12th, and 24th hours postoperatively. Pain scores will be evaluated at rest and during coughing using the Visual Analog Scale (VAS), where 0 = no pain and 10 = worst imaginable pain.
Total Postoperative Morphine Consumption | Within the first 24 hours after surgery
  Total morphine consumption in the first 24 hours after surgery will be recorded by the patient-controlled analgesia (PCA) device.

SECONDARY OUTCOMES:
Total Rescue Analgesic Use | Within the first 24 hours after surgery
  Amount of additional analgesic medication (excluding PCA-administered morphine) required in the first 24 hours postoperatively will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: murat izgi, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Only results
Supporting Information: Study Protocol, CSR
Time Frame: 2026-2030
Access Criteria: Individual participant data and supporting documents will be made publicly available without restriction

REFERENCES:
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Gagliese L, Katz J. Age differences in postoperative pain are scale dependent: a comparison of measures of pain intensity and quality in younger and older surgical patients. Pain. 2003 May;103(1-2):11-20. doi: 10.1016/s0304-3959(02)00327-5. PMID 12749954
- [Background] Sihoe ADL. Video-assisted thoracoscopic surgery as the gold standard for lung cancer surgery. Respirology. 2020 Nov;25 Suppl 2:49-60. doi: 10.1111/resp.13920. Epub 2020 Jul 30. PMID 32734596
- [Background] Feray S, Lubach J, Joshi GP, Bonnet F, Van de Velde M; PROSPECT Working Group *of the European Society of Regional Anaesthesia and Pain Therapy. PROSPECT guidelines for video-assisted thoracoscopic surgery: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2022 Mar;77(3):311-325. doi: 10.1111/anae.15609. Epub 2021 Nov 5. PMID 34739134
- See also: Link directs to a related article on the American Academy of Pain Medicine website, providing further details regarding the study's methodology and findings. — https://doi.org/10.5812/aapm-137664